CLINICAL TRIAL: NCT00360191
Title: A Placebo-Controlled Trial of Buspirone for Treatment of Marijuana Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: K23DA015440 (NIH); K23DA015440 (NIH)
Record Dates: First submitted 2006-08-02; First posted 2006-08-04 (Estimated); Last update posted 2012-01-12 (Estimated); Status verified 2007-12

CONDITIONS: Marijuana Abuse
MeSH Terms: conditions — Marijuana Abuse | interventions — Buspirone; Motivational Interviewing

INTERVENTIONS:
Drug: Buspirone
Procedure: Motivational enhancement therapy

SUMMARY:
The purpose of this study is to determine if buspirone combined with motivational enhancement therapy is effective in reducing marijuana use in marijuana-dependent adults.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy men and women, 18 years of age to 65 years of age.
2. Meet DSM-IV criteria for marijuana dependence.
3. All subjects will agree to and sign a written, IRB-approved informed consent.
4. Subjects must live within a 60-mile radius of Charleston, SC, in order to improve study visit compliance.
5. Subjects must be willing to identify collateral individuals for contact purposes to facilitate follow-up appointments.

Exclusion Criteria:

1. Individuals meeting DSM-IV dependence for a substance other than marijuana with the exception of nicotine and caffeine. Dependence on nicotine and caffeine will be allowed since dependence on these substances commonly co-occurs with marijuana dependence and excluding these individuals would compromise study recruitment.
2. Individuals meeting DSM-IV criteria for a lifetime history of schizophrenia or another non-affective psychotic disorder or bipolar disorder, since these patients will most likely be taking other psychotropic medications and often require intensive psychiatric care.
3. Individuals meeting DSM-IV criteria for current major depressive disorder or eating disorder, since these individuals will likely require treatment with psychotropic medications.
4. Individuals who present significant suicidal risk.
5. Individuals with significant cognitive impairment, as they may be unable to understand the informed consent, comply with study protocol, or accurately complete assessments.
6. Individuals currently receiving benzodiazepines, antidepressant or antipsychotic medications, as these medications could confound the effects of buspirone treatment.
7. Pregnant or nursing women, or women who refuse to use adequate birth control, as buspirone has not been approved for use in pregnancy.
8. Individuals without stable housing, as contacting these individuals would be difficult.
9. Individuals with major medical illnesses (e.g., HIV, renal failure, unstable angina, chronic obstructive pulmonary disease, infectious hepatitis).
10. Individuals who, in the investigators' opinion, would not be able to comply with study procedures, such as individuals unable to reliably present for intake appointments.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2004-04; Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aimee L McRae, PharmD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States